CLINICAL TRIAL: NCT01714440
Title: Genomics of Kidney Transplantation
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genomics of Transplantation Cooperative Research Program (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAIT GEN-03
Record Dates: First submitted 2012-10-17; First posted 2012-10-26 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: KidneyTransplant Recipients; Simultaneous Kidney/Pancreas Recipients; Kidney Transplant Donor
Keywords: genomics of kidney transplantation; genetic variation; recipient genotypes; donor genotypes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Transplant Recipients Cohort: Main Study Cohort: Kidney (or kidney-pancreas) transplant recipients. Enrollment for this cohort is closed.
- Transplant Donors Cohort: Main Study Cohort: The kidney donor for transplant recipients in this study. Enrollment for this cohort is closed.
- Activity&mRNA Expression Substudy Cohort: A subset of subjects enrolled in the main study who will receive tacrolimus, cyclosporine or mycophenolate as part of maintenance immunosuppression therapy. This group has a prospective observational cohort design. Enrollment into the Activity and messenger ribonucleic acid (mRNA) Expression Cohort, occurring concurrently with enrollment of the rest of the study, will continue until either the required sample size of 600 is achieved or the protocol team terminates enrollment. Participants in the Activity and mRNA Expression Cohort have additional blood draws up to 2 weeks prior to transplant, at week 1, Month 3 and Month 6 post-transplant.

SUMMARY:
The major aim of this research study is to investigate the relationship between genetic variation in DNA (inherited code material in the cells of the body) and factors affecting transplant outcomes, like the drugs people receive or the way their immune systems work, for example. To do this, investigators will collect blood samples from participants. Genetic material will be separated from each blood sample and analyzed, looking for genetic variation.

DETAILED DESCRIPTION:
In the past, the major problems in kidney transplantation were surgical complications, acute rejection, and infections. Right now, researchers are focusing on improving immune suppression therapy and achieving better long-term survival of kidney transplants. One of the ways to try to understand what causes loss of function after many years is to find out if there is a genetic factor involved.

There are a number of differences in specific genes that have been identified and are thought to affect transplant outcomes. Studying these gene variations (differences between people or differences between populations) is important in determining whether these variations are related to transplant outcomes and how this information can help patients achieve better long-term transplant survival.

ELIGIBILITY:
Inclusion Criteria:

* Kidney (or kidney-pancreas) transplant recipient no more than 10 days post-transplant or kidney donor no more than 30 days post-transplant or previously enrolled in Phase I of the Genomics of Kidney Transplantation Study;
* No organs other than kidney or pancreas transplanted simultaneously with the qualifying kidney transplant; and
* Participant or parent/guardian must be able to understand and provide written informed consent.

Inclusion for the Activity and mRNA Expression Cohort:

* Recipient enrolled in the Main Cohort Study;
* Informed consent for participation in the Activity and mRNA Expression Cohort;
* Age 18 years or greater as of day of transplantation;and
* Will receive tacrolimus, cyclosporine or mycophenolate as part of maintenance immunosuppression therapy.

Exclusion Criteria:

- Inability or unwillingness of the participant or parent/guardian to give a written informed consent or comply with the study protocol.

For the Activity and mRNA Expression Cohort:

- Inability or unwillingness of the participant or parent/guardian to give a written informed consent for participation in the Activity and mRNA Expression Cohort or comply with the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Targeted: 3000 Kidney or Kidney-pancreas transplant recipients and 1300 of the donors
Sampling Method: Non-Probability Sample
Enrollment: 1552 (Actual)
Dates: Start 2012-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Transplant recipient genotypes: time to chronic graft disfunction | Day 0 to Year 5
Transplant recipient genotypes: time to a persistent 25% decrease in Estimated Glomerular Filtration Rate (eGFR) | Day 0 to Year 5
  eGFR: Estimated GFR test results are a measure of kidney function.
Transplant recipient genotypes: time to acute rejection | Day 0 to Year 5
Transplant recipient genotypes: time to allograft failure | Day 0 to Year 5
  allograft failure is defined as graft loss or participant death.
Donor Genotypes: time to chronic graft dysfunction | Day 0 to Year 5
  The time to dysfunction of the donated organ.
Donor Genotypes: time to a persistent 25% decrease in eGFR | Day 0 to year 5
  The time to a persistent 25% decrease in eGFR in the donated organ's recipient.
Donor Genotypes: time to allograft failure | Day 0 to Year 5
  The time to the failure of the donated organ (defined as graft loss or participant death).
Recipient genotypes: time to select mycophenolate-related toxicities (leukopenia, anemia) | Day 0 to Year 5
Recipient genotypes: time to select Calcineurin Inhibitor (CNI)-related toxicities | Day 0 to Year 5
  Toxicities may include: new onset diabetes or nephrotoxicity. CNI: calcineurin inhibitor
Recipient genotypes: repeated measures of clinically obtained tacrolimus trough blood levels | Day 0 to Year 5
Recipient candidate genotypes: Calcineurin (CN) and IMPDH protein activity and expression | Day 0 to Year 5
  CN: Calcineurin. IMPDH: Inosine-5'-monophosphate dehydrogenase

SECONDARY OUTCOMES:
Time to composite endpoint of graft loss or death or persistent 25% increase in serum creatinine | Day 0 to Year 5
Time to renal biopsy with presence of the following semi-quantitative pathology endpoints: patterns of Banff biopsy score, presence of circulating anti-donor anti-Human Leukocyte Antigen (HLA) antibodies, C4d positivity | Day 0 to Year 5
Slope of eGFR | Day 0 to Year 5
Delayed graft function | Day 0 to Year 5
Time to Epstein-Barr virus (EBV) and Cytomegalovirus (CMV) infection | Day 0 to Year 5
  EBV: Epstein-Barr virus. CMV: cytomegalovirus.

CONTACTS AND LOCATIONS:
Overall Officials: A Matas, MD, Principal Investigator — University of Minnesota; A Israni, MD, MS, Study Chair — University of Minnesota
Locations (5):
- United States (4):
  - University of Alabama, Birmingham, Alabama
  - University of Minnesota, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Cao R, Schladt DP, Dorr C, Matas AJ, Oetting WS, Jacobson PA, Israni A, Chen J, Guan W. Polygenic risk score for acute rejection based on donor-recipient non-HLA genotype mismatch. PLoS One. 2024 May 31;19(5):e0303446. doi: 10.1371/journal.pone.0303446. eCollection 2024. PMID 38820342
- [Derived] Nguyen TT, Pearson RA, Mohamed ME, Schladt DP, Berglund D, Rivers Z, Skaar DJ, Wu B, Guan W, van Setten J, Keating BJ, Dorr C, Remmel RP, Matas AJ, Mannon RB, Israni AK, Oetting WS, Jacobson PA. Pharmacogenomics in kidney transplant recipients and potential for integration into practice. J Clin Pharm Ther. 2020 Dec;45(6):1457-1465. doi: 10.1111/jcpt.13223. Epub 2020 Jul 14. PMID 32662547
- [Derived] Oetting WS, Schladt DP, Dorr CR, Wu B, Guan W, Remmel RP, Ikle D, Mannon RB, Matas AJ, Israni AK, Jacobson PA; DeKAF Genomics and GEN03 Investigators. Analysis of 75 Candidate SNPs Associated With Acute Rejection in Kidney Transplant Recipients: Validation of rs2910164 in MicroRNA MIR146A. Transplantation. 2019 Aug;103(8):1591-1602. doi: 10.1097/TP.0000000000002659. PMID 30801535
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait